CLINICAL TRIAL: NCT03674463
Title: LCAR-B4822M-02 Cells in Treating Relapsed/Refractory (R/R) Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCAR-B4822M
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-09

CONDITIONS: Refractory or Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-B4822M treatment group (Experimental): r/r multiple myeloma patients will be treated with LCAR-B4822M CAR-T cells with a escalation approach, 0.5x10^6- 2.0x10^6 CAR-T cells/kg.
  Interventions: Drug: LCAR-B4822M CAR-T Cell Immunotherapy

INTERVENTIONS:
Drug: LCAR-B4822M CAR-T Cell Immunotherapy — Patients will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of CAR-T cells. After a pre-treatment lymphodepletion therapy, patients will receive the LCAR-B4822M CAR-T Cell Immunotherapy by intravenous injection.

SUMMARY:
This is a single arm, open-label, phase 1 study, to determine the safety and efficacy of LCAR-B4822M CAR-T cells in treating patients diagnosed with refractory/relapsed multiple myeloma (r/r MM).

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a usually incurable malignancy of plasma cells. Current therapies for multiple myeloma often cause remissions, but nearly all patients eventually relapse, there is an unmet clinical needs for these patients. B-cell maturation antigen (BCMA) is a protein expressed by normal plasma cells and the malignant plasma cells of multiple myeloma, and it was supposed to be a promising target for r/r MM.

ELIGIBILITY:
Inclusion Criteria:

- Patients must have a confirmed prior diagnosis of active multiple myeloma as defined by the updated IMWG criteria.

Patients with refractory multiple myeloma. Clear BCMA expression must be detected on malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry.

Refractory disease：1) At least 3 prior regimens, which must at least have contained bortezomi. or 2) other circumstances identified by clinical doctors.

Relapse criteria in NCCN clinical practice guidelines in Oncology: Multiple Myeloma (2016.V2)

Exclusion Criteria:

- Women of child-bearing potential or who are pregnant or breastfeeding. Have any active and uncontrolled infection: hepatitis B, hepatitis C, HIV, or other fatal viral and bacterial infection.

Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to either the required leukapheresis or the initiation of the conditioning chemotherapy regimen.

Patients with any uncontrolled intercurrent illness or serious uncontrolled medical disorder.

Patients with CNS metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions and spinal cord compression).

History of allogeneic stem cell transplantation. Have active acute or chronic graft-versus-host-disease (GVHD), or require immunosuppressant medications for GVHD, within 6 months of enrollment.

Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events | Day 1-30 days after injection
  Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Anti-myeloma responses to LCAR-B4822M cell treatment | Day 1-36 months after injection
  by measuring the changes of aberrant immunoglobulin in serum
Anti-myeloma responses to LCAR-B38M cell treatment | Day 1-36 months after injection
  multiple myeloma cells in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Hong Zhao, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided